CLINICAL TRIAL: NCT01479283
Title: Prophylactic Antibiotic Regimens in Tumor Surgery (PARITY): A Multi-Center International Randomized Controlled Trial Comparing Alternative Antibiotic Regimens in Patients Undergoing Tumor Resections With Endoprosthetic Replacements
Brief Title: Prophylactic Antibiotic Regimens in Tumor Surgery (PARITY)
Acronym: PARITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Orthopedic Research and Education Foundation (Other); The Physicians' Services Incorporated Foundation (Other); Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Michelle Ghert, MD, FRCSC, Professor | Department of Surgery, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GHRT01
Record Dates: First submitted 2011-11-15; First posted 2011-11-24 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Infection; Bone Neoplasms
Keywords: Infection; Bone Neoplasms; Prosthesis; Anti-Bacterial Agents; Randomized
MeSH Terms: conditions — Infections; Bone Neoplasms | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short-Arm Antibiotic Regimen (Active Comparator): Intervention: 24-Hour Prophylactic Cefazolin* Antibiotic Regimen
  *or another cephalosporin with equivalent gram-positive coverage in centers where cefazolin is not routinely used or not approved for use
  Interventions: Drug: 24-Hour Prophylactic Cefazolin* Antibiotic Regimen
- Long-Arm Antibiotic Regimen (Experimental): Intervention: 5-Days Prophylactic Cefazolin* Antibiotic Regimen
  *or another cephalosporin with equivalent gram-positive coverage in centers where cefazolin is not routinely used or not approved for use
  Interventions: Drug: 5-Days Prophylactic Cefazolin* Antibiotic Regimen

INTERVENTIONS:
Drug: 24-Hour Prophylactic Cefazolin* Antibiotic Regimen — Pre-Operative Antibiotic Regimen: Patients will receive 2g (or a weight-based dose based on 100mg/kg/day with a maximum single dose of 2g if < 18 years old) of IV cefazolin within 60 minutes prior to the procedure. No other pre-operative antibiotics will be administered.
  Intra-Operative Antibiotic Regimen: Patients will receive 2g (or a weight-based dose based on 100mg/kg/day with a maximum single dose of 2g if < 18 years old) of IV cefazolin every 3-4 hours. No other intra-operative antibiotics will be administered.
  Post-Operative Antibiotic Regimen: Patients will receive 2g (or a weight-based dose based on 100mg/kg/day with a maximum single dose of 2g if < 18 years old) of IV cefazolin every 8 hours for 24 hours followed by IV saline for 4 days. No other post-operative antibiotics will be administered.
  Other Names: ANCEF ®
  Arms: Short-Arm Antibiotic Regimen
Drug: 5-Days Prophylactic Cefazolin* Antibiotic Regimen — Pre-Operative Antibiotic Regimen: Patients will receive 2g (or a weight-based dose based on 100mg/kg/day with a maximum single dose of 2g if < 18 years old) of IV cefazolin within 60 minutes prior to the procedure. No other pre-operative antibiotics will be administered.
  Intra-Operative Antibiotic Regimen: Patients will receive 2g (or a weight-based dose based on 100mg/kg/day with a maximum single dose of 2g if < 18 years old) of IV cefazolin every 3-4 hours. No other intra-operative antibiotics will be administered.
  Post-Operative Antibiotic Regimen: Patients will receive 2g (or a weight-based dose based on 100mg/kg/day with a maximum single dose of 2g if < 18 years old) of IV cefazolin every 8 hours for 5 days. No other post-operative antibiotics will be administered.
  Other Names: ANCEF ®
  Arms: Long-Arm Antibiotic Regimen

SUMMARY:
The Prophylactic Antibiotic Regimens in Tumor Surgery (PARITY) trial is the first ever international multi-center randomized controlled trial in bone cancer surgery. In order to avoid amputation for bone cancer in the leg, complex limb-saving operations are performed. However, infections with devastating complications following surgery are common. Surgeons from across the world will randomize patients to receive either short- or long-duration antibiotic regimens after surgery with the goal of identifying the best regimen to reduce these infections.

DETAILED DESCRIPTION:
Long-bone sarcomas were historically managed with amputation. In the current era of osteosarcoma management, amputations are generally avoided by complex surgeries in which the malignancy is removed and the limb is reconstructed with advanced surgical techniques. This process of limb salvage is possible with improvements in chemotherapeutic regimens, advanced imaging techniques and surgical innovations such as modular metallic implants. However, the risk for surgical complications is high due to the complexity of the surgeries themselves. The most common and devastating complication is a surgical site infection. Background work and data from our pilot study indicates that infection rates approach 15%. Multiple surgical attempts at eradication of the infection fail in 50% of these cases, resulting in amputation. Published guidelines for post-operative antibiotic prophylaxis following many standard and less complex elective surgical procedures dictate that prophylactic antibiotics be discontinued after 24 hours. However, the most effective duration of treatment in sarcoma surgery has not previously been examined. Given the limitations of the evidence, it has not been possible for orthopaedic oncologists to draw firm conclusions and, therefore, clinical practice is highly varied, particularly with respect to antibiotic duration. Our international, multi-center randomized controlled trial will determine whether a 5-day regimen of post-operative prophylactic antibiotics in comparison to a standard 24-hour regimen decreases the rate of surgical site infections after limb salvage surgery within 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* primary bone malignancies or aggressive benign bone tumors of the femur or tibia, soft-tissue sarcomas which have invaded the femur or tibia, or oligometastatic bone disease of the femur or tibia in a patient expected to live at least one year post-operatively; and
* treatment by surgical excision and endoprosthetic replacement of the femur or tibia.

Exclusion Criteria:

* current known Methicillin-resistant Staphylococcus Aureus (MRSA) colonization;
* current known Vancomycin Resistant Enterococcus (VRE) colonization;
* documented anaphylaxis or angioedema to penicillin or cefazolin (Ancef);
* current surgical procedure is a revision surgery for implant failure or infection;
* prior local infection within the surgical field of the affected limb;
* current known immunologically-deficient disease conditions (not including recent chemotherapy);
* known renal insufficiency with estimated creatinine clearance (eGRF) of less than 54 mL/min;
* reconstruction to include structural allograft;
* enrolled in a competing study; and
* weight of less than or equal to 45 kg (for sites using cefuroxime only).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infections | 1 year
  the development of a surgical site infection according to the criteria established by the Center for Disease Control (CDC)

SECONDARY OUTCOMES:
Functional Outcome and Quality of Life | 1 year
  as measured by the Musculoskeletal Tumor Society (MSTS) functional score (1987 and 1993 versions) and the Toronto Extremity Salvage Score (TESS) questionnaires
Antibiotic-Related Complications | 1 year
  examples of antibiotic-related complications include gastrointestinal infections, fungal infections, etc.
Rate of Re-Operation | 1 year
  re-operation may be required if patients develop a surgical site infection
Oncologic Recurrence and/or Metastases | 1 year
Mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Ghert, MD, FRCSC, Principal Investigator — McMaster University
Locations (54):
- United States (34):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford University Hospital and Clinics, Redwood City, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Francisco Medical Center, San Francisco, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Emory Orthopaedics and Spine Center, Atlanta, Georgia
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Franklin Square Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - SUNY Upstate University Hospital, East Syracuse, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Long Island Jewish Medical Center | Northwell Health, Queens, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Cleveland Clinic - Hillcrest Hospital, Cleveland, Ohio
  - Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - The Rothman Institute at Jefferson, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Hospital Universitario Austral, Pilar, Buenos Aires, Argentina
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- LKH - Universitätsklinikum Graz, Graz, Austria
- Brazil (2):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Instituto de Ortopedia e Traumatologia, São Paulo
- Canada (8):
  - Foothills Medical Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hôtel-Dieu de Québec, Québec, Quebec
- Children's Cancer Hospital Egypt, Cairo, Egypt
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - University Medical Center Groningen, Groningen
- Singapore General Hospital, Singapore, Singapore
- Grey's Hospital, Pietermaritzburg, South Africa
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hasan K, Racano A, Deheshi B, Farrokhyar F, Wunder J, Ferguson P, Holt G, Schwartz H, Petrisor B, Bhandari M, Ghert M. Prophylactic antibiotic regimens in tumor surgery (PARITY) survey. BMC Musculoskelet Disord. 2012 Jun 7;13:91. doi: 10.1186/1471-2474-13-91. PMID 22676321
- [Background] Ghert M, Deheshi B, Holt G, Randall RL, Ferguson P, Wunder J, Turcotte R, Werier J, Clarkson P, Damron T, Benevenia J, Anderson M, Gebhardt M, Isler M, Mottard S, Healey J, Evaniew N, Racano A, Sprague S, Swinton M, Bryant D, Thabane L, Guyatt G, Bhandari M; PARITY Investigators. Prophylactic antibiotic regimens in tumour surgery (PARITY): protocol for a multicentre randomised controlled study. BMJ Open. 2012 Nov 28;2(6):e002197. doi: 10.1136/bmjopen-2012-002197. Print 2012. PMID 23194956
- [Background] Racano A, Pazionis T, Farrokhyar F, Deheshi B, Ghert M. High infection rate outcomes in long-bone tumor surgery with endoprosthetic reconstruction in adults: a systematic review. Clin Orthop Relat Res. 2013 Jun;471(6):2017-27. doi: 10.1007/s11999-013-2842-9. Epub 2013 Feb 12. PMID 23404421
- [Background] Evaniew N, Nuttall J, Farrokhyar F, Bhandari M, Ghert M. What are the levels of evidence on which we base decisions for surgical management of lower extremity bone tumors? Clin Orthop Relat Res. 2014 Jan;472(1):8-15. doi: 10.1007/s11999-013-3311-1. Epub 2013 Oct 1. PMID 24081669
- [Derived] Prophylactic Antibiotic Regimens in Tumor Surgery (PARITY) Investigators; Ghert M, Schneider P, Guyatt G, Thabane L, Velez R, O'Shea T, Randall RL, Turcotte R, Wilson D, Wunder JS, Baptista AM, Cheng EY, Doung YC, Ferguson PC, Giglio V, Hayden J, Heels-Ansdell D, Khan SA, Sampath Kumar V, McKay P, Miller B, van de Sande M, Zumarraga JP, Bhandari M. Comparison of Prophylactic Intravenous Antibiotic Regimens After Endoprosthetic Reconstruction for Lower Extremity Bone Tumors: A Randomized Clinical Trial. JAMA Oncol. 2022 Mar 1;8(3):345-353. doi: 10.1001/jamaoncol.2021.6628. PMID 34989778
- [Derived] Schneider P, Heels-Ansdell D, Thabane L, Ghert M; PARITY Investigators. Prophylactic Antibiotic Regimens In Tumor Surgery (PARITY): a multi-center randomized controlled study comparing alternative antibiotic regimens in patients undergoing tumor resections with endoprosthetic replacements-a statistical analysis plan. Trials. 2021 Mar 22;22(1):223. doi: 10.1186/s13063-021-05147-2. PMID 33752752
- [Derived] Gazendam A, Bozzo A, Schneider P, Giglio V, Wilson D, Ghert M. Recruitment patterns in a large international randomized controlled trial of perioperative care in cancer patients. Trials. 2021 Mar 20;22(1):219. doi: 10.1186/s13063-021-05149-0. PMID 33743753